CLINICAL TRIAL: NCT06628635
Title: Examining the Effects of Aerobic Exercise, Isometrics, and Stretching on Acute (Post-exercise) Blood Pressure Reduction
Brief Title: Examining Different Modes of Exercise for Acute Reduction in Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Phil Chilibeck, Professor, University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023_24_09
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Hypertension
Keywords: blood pressure; exercise
MeSH Terms: conditions — Hypertension; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Aerobic exercise (Experimental): 30 minutes of moderate-intensity aerobic exercise on a cycle ergometer
  Interventions: Behavioral: Exercise
- Isometric exercise (Experimental): 30 minutes of isometric exercise (alternating hand-grip with wall-sitting)
  Interventions: Behavioral: Exercise
- Static stretching (Experimental): 30 minutes of static stretching of major muscle groups
  Interventions: Behavioral: Exercise
- Resting control (Active Comparator): 30 minutes of seated rest
  Interventions: Behavioral: Resting

INTERVENTIONS:
Behavioral: Exercise — Exercise involving aerobics, isometrics, and stretching
  Arms: Aerobic exercise; Isometric exercise; Static stretching
Behavioral: Resting — Resting
  Arms: Resting control

SUMMARY:
The purpose of the study is to compared different modes of exercise for eliciting post-exercise hypotension. The study will randomize 10 healthy participants to 30 minutes of either aerobic exercise, isometric exercise, stretching, or rest (control). Blood pressure and heart rate will be assessed before and for one hour post-exercise.

DETAILED DESCRIPTION:
The purpose is to compare different modes of exercise (aerobic vs. isometric vs. static stretching) for reducing blood pressure post-exercise. : Using a randomized crossover design, 5 male and 5 female (n=10) normotensive university students will participate in four different exercise sessions for 30 minutes: aerobic (cycle ergometer at 70% of VO2max), isometric (alternating wall-sit for 70% of max, and handgrip dynamometer at 30% of max for 2 minutes), stretching (targeting the larger muscle groups of the body), and control (rest). Participants' blood pressure and heart rate will be measured before each exercise session and monitored for 60 minutes afterwards to analyze the post-exercise hypotensive response.

ELIGIBILITY:
Inclusion Criteria:

* Able to safely perform exercise according to the Get Active Questionnaire

Exclusion Criteria:

* Taking blood pressure medications

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-01-04 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Change in systolic blood pressure (mmHg) | Baseline to 60 minutes after exercise
Change in diastolic blood pressure (mmHg) | Baseline to 60 minutes after exercise

SECONDARY OUTCOMES:
Change in heart rate (beats per minute) | Baseline to 60 minutes after exercise
Change in rate-pressure product (beats per mintues x systolic blood pressure mmHg) | Change from baseline to 60 minutes after exercise

CONTACTS AND LOCATIONS:
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Keller C, Chilibeck P. Stretching, isometrics, and aerobic exercise for decreasing blood pressure post-exercise: a randomized crossover study. Appl Physiol Nutr Metab. 2025 Jan 1;50:1-6. doi: 10.1139/apnm-2024-0439. PMID 39869856